CLINICAL TRIAL: NCT06813456
Title: Implementation of Solid Digital PCR to Support Gold-standard Methods for Evaluation of HER2 Amplification Status: Focus on HER2-low Subtype
Acronym: CRANBERRY
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CRANBERRY; RC-2024-2790620 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2024-12-09; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; HER2; HER2-low; Prognostic-predictive markers; IHC; D-DISH; FISH; solid digital PCR; liquid biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — FFPE, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of the retrospective phase of this study is to validate the specificity and the sensitivity of two Real-Time quantitative PCR based techniques in order to support the gold-standard approaches used to evaluate the HER2 gene status in breast cancer.

Furthemore, HER2-low patients are enrolled in a prospective phase, both in early stage and in case of recurrence, in order to monitorate HER2 expression levels changes under treatments by using liquid biopsy. The first aim is to be able to distinguish responders vs non-responders earlier than the standard monitoring through tumoral markers and medical examination.

DETAILED DESCRIPTION:
The hypothesis underlying this study is that the use of solid digital PCR technology and the MammaTyper® diagnostic test allows the molecular classification of breast carcinomas to be refined and strengthened from early diagnosis, limiting the bias related to interpretation problems and thus improving the prognostic power of traditional clinical pathological parameters. In fact, the quantitative data of each individual marker, associated with the molecular subtype, provides the oncologist with indispensable prognostic information to define the most appropriate therapeutic approach.

Specifically, it is believed that the use of more accurate methods to define HER2 amplification status may help improve diagnostic accuracy, as well as support the choice of optimal therapy, especially for the new HER2-low tumour subtype.

It is believed that HER2 levels defined in this way, once correlated with clinical data on survival and response to the therapeutic regimen undertaken by each patient, will allow the detection of significant differences between the HER2-positive, -negative and -equivocal groups, the latter needing to be reclassified as separate entities.

A further hypothesis concerns the possible impact that dPCR technology may have in predicting and monitoring response to therapies in a robust, rapid and cost-effective manner. The first endpoint of this study is the identification, by quantitative analysis with dPCR and Mammatyper® performed on paraffin-embedded archival tissue, of HER2-amplified and -unamplified breast carcinomas, the expression levels of which will be compared with those detected by gold-standard methods in order to resolve cases that are difficult to interpret. With the molecular test Mammatyper® it will also be possible to objectively and reproducibly determine the expression of the prognostic-predictive markers ER, PR and Ki67. It is expected that the clinical outcomes of patients will correlate significantly with the expression levels of ER, PR, Ki67 and HER2 estimated in the study.

The second endpoint of the study is the identification, by quantitative dPCR analysis performed on paraffin-embedded tissue and liquid biopsy, of HER2-0 and HER2-low enrolled early-stage breast carcinomas undergoing surgical and systemic therapy.It is expected to detect any fluctuations in HER2 expression/amplification due to sensitivity/resistance to systemic therapy or, at follow-up, recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologic confirmation of breast cancer from 1/1/2022
* Patient treated with systemic and surgical therapy (retrospective phase)
* Signed informed consent
* HER2-0 and/or HER2-low patient, according to IHC and D-DISH/FISH, treatable with systemic and surgical therapy (prospective phase)

Exclusion Criteria:

* Lack of molecular classification on the basis of prognostic-predictive markers ER, PR, Ki67 and HER2 (Luminal A, Luminal B HER2-positive, Luminal B HER2- negative, HER2-positive, Triple negative)
* Prior neoplasms, other than the neoplasm under investigation, arised within the past 5 years
* Missing histological diagnosis of HER2-0 and/or HER2-low breast cancer (prospective phase)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population considered for the retrospective phase of the study will consist of women with stage I-III breast cancer, aged 18 years and older, who have accessed the SSD of Breast Surgery and Oncology of IRCCS - Azienda Ospedaliero-Universitaria di Bologna Policlinico di S.Orsola, in the context of the normal care path provided for patients with this pathology (first histopathological diagnosis from 1/1/2022).
  The population considered for the prospective phase of the study will consist of women with early-stage HER2-0 and HER2-low breast cancer (population 1) or metastatic HER2-low breast cancer (population 2), 18 years of age and older, who will be referred to the SSD of Breast Surgery and Oncology of IRCCS - Azienda Ospedaliero-Universitaria di Bologna Policlinico di S.Orsola.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Breast cancer patients undergone surgical and systemic therapy | At baseline
  Estimation of sensitivity and specificity confidence intervals of MammaTyper and dPCR threshold values in discriminating HER2 positivity on FFPE tissues and comparison with gold-standard approaches.
Early-stage HER2-low breast cancer patients undergoing surgical and systemic therapy | At baseline
  Sensitivity and specificity of HER2 expression values according to dPCR performed on FFPE tissue and according to dPCR performed on liquid biopsy, compared with the gold-standard approaches
Metastatic HER2-low patients in treatment with Trastuzumab-Deruxtecan | Every 4 months from the start of therapy,assessed up to 60 months
  Response to Trastuzumab-Deruxtecan therapy to be assessed by tumor markers, radiological investigations and clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Coluccelli, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No